CLINICAL TRIAL: NCT04105387
Title: Timing of First Tracheostomy Change
Brief Title: Tracheostomy Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-014348
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Tracheostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Tracheostomy change at day 7
- Treatment Group (Experimental): Tracheostomy change at day 4
  Interventions: Procedure: Early Tracheostomy Change

INTERVENTIONS:
Procedure: Early Tracheostomy Change — The treatment group will have the first tracheostomy change on postoperative day 4 by an Otolaryngology physician (attending or fellow) on the study team.
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to compare outcomes of first tracheostomy change on postoperative day 4 to our current standard of care of first tracheostomy change on postoperative day 7.

DETAILED DESCRIPTION:
A "fresh tracheostomy" is a tracheostomy whose tract is not yet well formed and that has not yet been changed since the operative procedure. It is considered a "critical airway" since replacement following dislodgement may be difficult and at risk of forming a false tract. Thus, an infant or a child with a fresh tracheostomy is cared for in the intensive care unit and kept sedated to prevent accidental dislodgement. During this time wound care is often suboptimal due to fear of manipulating the neck. Patients are at increased risk of complications such as pressure ulcers and pneumonia related to being sedated for an extended length of time. Furthermore, prolonged sedation can lead to difficulties with withdrawal and delay recovery. Progression of the patient's care and the teaching of tracheostomy care to caregivers is also delayed. Thus, timing of the first tracheostomy change has great implications for prevention of complications as well as length of hospital stay. While in adults is it accepted that the first trach change can be done as early as post-operative day 3. In pediatrics no good evidence or clear guidelines is available as to when the first tracheostomy change should occur. It is common to wait until days 5-7 which allows establishment of a mature tract however, there is no biologic reason to think that a pediatric tracheostomy tract should take any longer to epithelize than in an adult. Several studies have reported safe tracheostomy change in pediatric patients as early as postoperative day 3 (Deutsch 1998, Lippert 2014, Van Buran 2014). Currently at CHOP our standard of care is to perform the first tracheostomy change on post-operative day 7. The investigators aim to compare tracheostomy tube change at post-operative day 4 by randomizing patients undergoing tracheostomy at CHOP to day 4 (treatment) or day 7 (control) groups.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 0 to 2 years of age at the time of tracheostomy.
2. Scheduled to undergo tracheostomy, or underwent tracheostomy and is currently postoperative day 4 or less
3. Parental/guardian permission (informed consent)

Exclusion Criteria:

1. Anatomical or physiological states identified preoperatively or intraoperatively that, in the investigator's judgment, raise concern over the viability of the tracheostomy tract to form within the first several days, or would otherwise increase the difficulty of performing an early tracheostomy change.
2. Previous or concomitant surgery at tracheostomy site
3. Subjects who cannot be physically intubated orally or for whom intubation would be difficult for the experienced ears nose and throat physician
4. Subjects who cannot be mask ventilated

Subjects that do not meet all of the enrollment criteria may not be enrolled. Any violations of these criteria must be reported in accordance with Institutional Review Board Policies and Procedures.

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Difference in complication rates between tracheostomy change group subjects | 6 weeks
  This will be evaluated by analyzing a difference in proportions between the "day 4" group and "day 7" group for tracheostomy changes. This will be analyzed during the study participation, regardless of which group the subjects belong to. The analysis will be conducted using two-samples tests for difference in proportions between two study groups, using a two-sided chi-square test at significance level of 0.05.

SECONDARY OUTCOMES:
The difference in length of ICU stay between change group subjects | 6 weeks
  The analyses will use two-sample t-test or Mann-Whitney (as appropriate) test to compare the length of ICU/hospital stay between "day 4" group and "day 7" group subjects. This will be analyzed during the study participation, regardless of which group the subjects belong to.
The difference in duration of sedation between change group subjects | 6 weeks
  The analyses will use two-sample t-test or Mann-Whitney (as appropriate) test to compare the duration of sedation between "day 4" group and "day 7" group subjects. This will be analyzed during the study participation, regardless of which group the subjects belong to.
The difference in the amount of time for parent/caregiver education between change subjects | 6 weeks
  The analyses will use two-sample t-test or Mann-Whitney (as appropriate) test to compare the the amount of time for parent/caregiver education between "day 4" group and "day 7" group subjects. This will be analyzed during the study participation, regardless of which group the subjects belong to.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deutsch ES. Early tracheostomy tube change in children. Arch Otolaryngol Head Neck Surg. 1998 Nov;124(11):1237-8. doi: 10.1001/archotol.124.11.1237. PMID 9821926
- [Background] Lippert D, Hoffman MR, Dang P, McMurray JS, Heatley D, Kille T. Care of pediatric tracheostomy in the immediate postoperative period and timing of first tube change. Int J Pediatr Otorhinolaryngol. 2014 Dec;78(12):2281-5. doi: 10.1016/j.ijporl.2014.10.034. Epub 2014 Nov 3. PMID 25468464
- [Background] McCullagh, Peter; Nelder, John. Generalized Linear Models, Second Edition 1989. Boca Raton: Chapman and Hall/CRC.
- [Background] McEvoy TP, Seim NB, Aljasser A, Elmaraghy CA, Ruth B, Justice L, Begue S, Jatana KR. Prevention of post-operative pediatric tracheotomy wounds: A multidisciplinary team approach. Int J Pediatr Otorhinolaryngol. 2017 Jun;97:235-239. doi: 10.1016/j.ijporl.2017.03.037. Epub 2017 Mar 31. PMID 28483242
- [Background] Mitchell RB, Hussey HM, Setzen G, Jacobs IN, Nussenbaum B, Dawson C, Brown CA 3rd, Brandt C, Deakins K, Hartnick C, Merati A. Clinical consensus statement: tracheostomy care. Otolaryngol Head Neck Surg. 2013 Jan;148(1):6-20. doi: 10.1177/0194599812460376. Epub 2012 Sep 18. PMID 22990518
- [Background] Senders CW, Muntz HR, Schweiss D. Physician survey on the care of children with tracheotomy. Am J Otolaryngol. 1991 Jan-Feb;12(1):48-50. doi: 10.1016/0196-0709(91)90072-n. PMID 2029066
- [Background] Van Buren NC, Narasimhan ER, Curtis JL, Muntz HR, Meier JD. Pediatric tracheostomy: timing of the first tube change. Ann Otol Rhinol Laryngol. 2015 May;124(5):374-7. doi: 10.1177/0003489414560430. Epub 2014 Nov 27. PMID 25432165